CLINICAL TRIAL: NCT00313963
Title: MAST - Magnesium for Sickle Cell Acute Crisis in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000008367
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Anemia, Sickle Cell
Keywords: Anemia, Sickle Cell; Magnesium Sulfate; pediatric
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Magnesium Sulfate
- 2 (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — Intravenous Magnesium Sulfate (100 mg/Kg, Max 2 gram/dose) 8 hourly.
  Arms: 1
Drug: Normal Saline — Intravenous Placebo (Normal Saline in equivalent amount to magnesium sulfate 100 mg/Kg, Max 2 gram/dose) 8 hourly.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if intravenous magnesium sulfate treatment is effective in reducing the length of stay and pain in children with sickle cell disease suffering an acute vaso-occlusive episode.

DETAILED DESCRIPTION:
Sickle cell disease is a group of complex, chronic disorders characterized by hemolysis, acute vaso-occlusive episodes (crises), unpredictable acute complications that can be life-threatening, and the variable development of chronic organ damage. Administration of magnesium sulfate has the potential to reduce hemolysis since it induces negatively charged chloride ions and water entry to the cell. To date only one non-randomized, non-blinded, single arm study with only 19 children evaluated the effect of magnesium on length of stay in the hospital of children with sickle cell disease.

In this randomized, double blind, two-arm placebo controlled study, children with sickle cell disease admitted for a vaso-occlusive crisis will receive intravenous magnesium sulfate or placebo every 8 hours during their stay in the hospital , along with pain management. We will measure length of stay (LOS), pain, adverse effects, and the total amount of narcotics required for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Known sickle cell disease
* Previous painful crisis resulting in an Emergency Department(ED) visit
* Current visit with a chief complaint of pain
* Age 4 years - 18 years
* Staff ED decides to admit to the hospital
* Staff ED decides to start an intravenous line

Exclusion Criteria:

* Fever (>38.5C) during the 24 hours prior to visit at triage
* Patients transfused within 90 days of study entry
* Patients with known renal disease
* Patients with known heart block or myocardial damage
* Patients who take a magnesium-containing medication or calcium channel blocker on a regular basis
* Patients who received anesthetics, cardiac glycosides and neuromuscular blockers during the acute illness in the last 24 hours
* Patients or parents unable to communicate in English
* Known pregnancy
* Known allergy to Magnesium
* Admission to the ICU
* Enrolment to the study in the last 30 days

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2006-04; Primary Completion 2008-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Length of stay in the hospital | Time frame determined by outcome

SECONDARY OUTCOMES:
Reduction mean daily pain score during an admission for sickle cell pain crisis | Length of hospital stay
Adverse events during admission | Length of hospital stay
Cumulative Narcotic drug required to manage the crises during admission | Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Friedman, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Goldman RD, Mounstephen W, Kirby-Allen M, Friedman JN. Intravenous magnesium sulfate for vaso-occlusive episodes in sickle cell disease. Pediatrics. 2013 Dec;132(6):e1634-41. doi: 10.1542/peds.2013-2065. Epub 2013 Nov 25. PMID 24276838